CLINICAL TRIAL: NCT02558205
Title: Establishing a Correlation Between Pre-treatment CT Perfusion Parameter Values and Post-treatment PET/CT Dosimetry to Aid in Tumor-specific Y-90 Radioembolization Treatment Planning for Hepatocellular Carcinoma
Brief Title: Correlation Between CT Perfusion and Post Y-90 TARE PET/CT Dosimetry
Status: Withdrawn | Type: Observational
Why Stopped: unable to rectuir
Sponsor: Rush University Medical Center (Other)
Collaborators: Swim Across America (Other)
Responsible Party: Sponsor
Other Study IDs: 14100902
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CT Perfusion and PET/CT: Patients undergo both a CT liver perfusion study pre Y-90 treatment and a PET/CT of liver following Y-90 treatment. For the PET/CT no additional radioactivity is required.
  Interventions: Radiation: CT Liver Perfusion; Radiation: PET/CT of liver

INTERVENTIONS:
Radiation: CT Liver Perfusion — Imaging study of liver using injection of Iodine contrast agent done using CT imaging
Radiation: PET/CT of liver — PET/CT of liver following Y-90 treatment. PET/CT imaging uses positron decay of Y-90 to detect distribution of Y-90 in the liver.

SUMMARY:
The purpose of this study is to see if it is possible to establish a relationship between the blood flow and blood volume of liver tumors from CT body perfusion and the radiation dose deposited in the tumors from the radioembolization treatment as measured by PET/CT.

The study will do this by:

1. Measuring the blood flow and blood volume of tumors in the imaging data from a CT body perfusion
2. Measuring the radioactivity in the tumors after the radioembolization treatment using PET/CT and then calculating the dose deposited in the tumor
3. Using statistical analysis to assess the relationship between the dose and the perfusion parameters

In addition, the research may help develop a method for calculating the dose of radioembolization to be delivered to a liver tumor(s) using blood volume and blood flow data obtained from the CT body perfusion scans.

DETAILED DESCRIPTION:
The overreaching goal of this line of research is to establish a methodology to produce patient and tumor specific treatment planning for Yttrium-90 radioembolization of hepatocellular carcinoma (HCC). The proposed project will facilitate the collection of preliminary data to support a larger study to more fully establish the relationship between tumor perfusion parameters and delivered radiation dose. Y-90 radioembolization delivers millions of small resin or glass beads attached to or containing (depending on the product) the beta emitting radioisotope of Yttrium. These beads are injected into the patient's hepatic artery during an interventional radiology procedure. The beads are pushed into the hepatic vasculature system by pulsatile flow and eventually become lodged, due to their finite size, in the microvasculature of the liver and tumor and deliver the radiation dose from the high energy beta particles (average energy 0.94 MeV) released during the radioactive decay (half life of 64 hours) in a highly local (~2.5 mm range) manner. The beads are permanently embedded in the vasculature and the radioactivity eventually decays to background.

Current practice is to calculate and deliver an average liver lobe radiation dose based on either the lobar volume or the patient's body surface area. However, because of the hypervascular nature of HCC lesions, the tumors receive a greater proportion of the beads than the healthy liver parenchyma and hence are assumed to receive radiation doses well above that of calculated average liver dose and the dose to the normal liver. Due to the differing vascularity and characteristics of tumors and patients, each Y-90 treatment does not deliver the same dose to the tumor. A less vascular tumor may receive substantially less radiation than a more vascular one which affects the tumoricidal efficacy of the treatment and ultimately the patient's final outcome. New techniques using Positron Emission Tomography (PET)/CT following Y-90 treatment allow for retrospective dosimetry to determine the actual dose delivered to the tumor. However, no methodology exists to plan the dose to be delivered to the tumor prior to the treatment.

This research aims to collect preliminary data to begin to establish a prospective method to use Computed Tomography (CT) perfusion studies of the liver to calculate the expected dose to the HCC lesions and the normal liver based on the blood flow and blood volume. This goal will be achieved by prospectively collecting CT Perfusion studies prior to Y-90 radioembolization treatments and PET/CT immediately following treatments. The relationship between the perfusion parameters representing the vascularity of the lesions and the normal liver and the post treatment PET/CT dosimetry will be established by this line of research. The hypothesized correlation between the perfusion parameters and the tumor dose as established by PET/CT will allow for patient and tumor specific treatment planning ensuring that the appropriate tumoricidal radiation dose is reliably delivered.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular Carcinoma diagnosis
* Candidate for Trans-Arterial Radioembolization treatment

Exclusion Criteria:

* Less than 18 years old
* Pregnant
* Iodinated Contrast Agent Allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified for Y-90 transarterial radioembolization of liver tumors with hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of CT perfusion metrics to radiation dose deposition of Y-90 as measured by PET/CT | 1 year

SECONDARY OUTCOMES:
Correlation between CT perfusion metrics and post treatment response as measured by RECIST 1.0 criteria | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Supanich, Ph.D., Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Frampas E, Lassau N, Zappa M, Vullierme MP, Koscielny S, Vilgrain V. Advanced Hepatocellular Carcinoma: early evaluation of response to targeted therapy and prognostic value of Perfusion CT and Dynamic Contrast Enhanced-Ultrasound. Preliminary results. Eur J Radiol. 2013 May;82(5):e205-11. doi: 10.1016/j.ejrad.2012.12.004. Epub 2012 Dec 28. PMID 23273822
- [Background] Morsbach F, Sah BR, Spring L, Puippe G, Gordic S, Seifert B, Schaefer N, Pfammatter T, Alkadhi H, Reiner CS. Perfusion CT best predicts outcome after radioembolization of liver metastases: a comparison of radionuclide and CT imaging techniques. Eur Radiol. 2014 Jul;24(7):1455-65. doi: 10.1007/s00330-014-3180-3. Epub 2014 May 12. PMID 24817083
- [Background] Lea WB, Tapp KN, Tann M, Hutchins GD, Fletcher JW, Johnson MS. Microsphere localization and dose quantification using positron emission tomography/CT following hepatic intraarterial radioembolization with yttrium-90 in patients with advanced hepatocellular carcinoma. J Vasc Interv Radiol. 2014 Oct;25(10):1595-603. doi: 10.1016/j.jvir.2014.06.028. Epub 2014 Aug 23. PMID 25156647
- [Background] Bourgeois AC, Chang TT, Bradley YC, Acuff SN, Pasciak AS. Intraprocedural yttrium-90 positron emission tomography/CT for treatment optimization of yttrium-90 radioembolization. J Vasc Interv Radiol. 2014 Feb;25(2):271-5. doi: 10.1016/j.jvir.2013.11.004. PMID 24461132
- [Background] D'Arienzo M, Filippi L, Chiaramida P, Chiacchiararelli L, Cianni R, Salvatori R, Scopinaro F, Bagni O. Absorbed dose to lesion and clinical outcome after liver radioembolization with 90Y microspheres: a case report of PET-based dosimetry. Ann Nucl Med. 2013 Aug;27(7):676-80. doi: 10.1007/s12149-013-0726-4. Epub 2013 Apr 20. PMID 23605058